CLINICAL TRIAL: NCT01313611
Title: BRIEF: Bendamustine and Rituximab In Elderly Follicular: A Multicentric Phase II Study Evaluating the Benefit of a Short Induction Treatment by Bendamustine and Rituximab Followed by Maintenance Therapy With Rituximab In Elderly (≥ 60 Years Old) Patients With Untreated Follicular Lymphoma Patients, With an Intermediate or High FLIPI Score
Brief Title: BRIEF Bendamustine and Rituximab In Elderly Follicular
Acronym: BRIEF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treament with rituximab during maintenance phase was stoped, according to DSMC recommendations, since 3 cases of deaths occured.
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRIEF
Record Dates: First submitted 2011-02-21; First posted 2011-03-14 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab + bendamustine (Experimental)
  Interventions: Drug: Rituximab + bendamustine

INTERVENTIONS:
Drug: Rituximab + bendamustine — Induction phase: rituximab and bendamustine on Day 1, Bendamustine on Day 2, Rituximab on Day 8, Rituximab on Day 15, Rituximab on Day 22, bendamustine on Day 29, Bendamustine on Day 30

SUMMARY:
The objective of this study is to evaluate the complete response rate after a short induction treatment with rituximab (375mg/m2)and bendamustine (90mg/m2)in In Elderly (≥ 60 years old) patients with untreated Follicular lymphoma, with an intermediate or high FLIPI score and without high tumor burden.

This short induction is followed by a rituximab (375mg/m2)maintenance/ Induction schedule:Rituximab+Bendamustine on Day 1, Bendamustine on Day 2, Rituximab on Day 8, Rituximab on Day 15, rituximab on day 22, Bendamustine on Day 29, Bendamustine on Day 30 Maintenance schedule: 12 infusions of rituximab, each 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma CD20+, all grades except the grade 3b with a lymph node biopsy performed within 6 months before study entry and with material available for central review
* A minimal initial immunology is required, including : CD20, bcl-2, CD10 and CD5
* Age must be ≥ 60 years
* Patients not previously treated
* Patients with an intermediate or high risk FLIPI score requiring 2 or more of the following adverse prognostic factors:

  1. Age >60 ans
  2. Ann Arbor Stage (III-IV vs. I-II)
  3. Hemoglobin level ( < 12g/dL vs. ≥ 12 g/dL)
  4. Number of nodal areas (< 5 vs. ≥ 5) (Note: LDH should not be considered as an adverse prognostic factor in this study since it is considered as high tumor burden in the GELF criteria)
* Low burden disease at study entry according to the GELF criteria
* Patients with at least one measurable site of disease: patients with only blood or marrow or splenic infiltration are excluded
* Performance status ≤ 2 on the ECOG scale
* Adequate hematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow) including:
* Hemoglobin ≥ 8.0 g/dL (5.0 mmol/L)
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Adequate renal function: calculated creatinine clearance > 50 ml/min (according to MDRD method) unless these abnormalities are related to lymphoma
* Adequate hepatic function: Total bilirubin < 2.0 mg/dl (34 µmol/L), AST (SGOT) and ALT (SGPT) ≤ 2.5 x the upper limit of normal unless these abnormalities are related to lymphoma
* Adequate cardiac function: LEVF ≥ 50% calculated by echocardiography or scintigraphy
* Having previously signed a written informed consent

Exclusion Criteria:

* Other histological types of lymphoma than follicular lymphoma
* Grade 3b follicular lymphoma
* Patients previously on watch and wait since more than 6 months from diagnosis
* Patients previously treated for lymphoma, except splenectomy
* Patients with low FLIPI score (0 or 1 adverse prognostic factors not considering elevated LDH)
* Bulky disease at study entry according to the GELF criteria
* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningitis)
* Patients with prior or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer or previous cancer in CR without any treatment in the last 5 years
* Positive HIV, HBV (anti-HBc positivity) and HCV serologies before inclusion
* Poor Performance status > 2 on the ECOG scale
* Known contra-indication to study product
* Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease).
* Any other co-existing medical or psychological condition that will preclude participation in the study or compromise ability to give informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Complete response rate according to Cheson criteria 1999 after a short induction treatment by rituximab and bendamustine | 12 weeks

SECONDARY OUTCOMES:
Complete response rate according to Cheson criteria 1999 after 24 months of maintenance therapy with Rituximab | 26 months
Partial and objective response rates at the end of induction phase | 12 weeks
Duration of response | From the time of attainment of CR or PR to the date of first documented disease progression, relapse or death from any cause
Progression free survival | From the date of randomization to the date of first documented disease progression, relapse, initiation of new anti-lymphoma therapy or death from any cause.
Overall survival | From the date of randomization to the date of death from any cause
Time before retreatment | From the end of primary treatment until the institution of the next therapy
Immediate toxicity | 12 weeks
Long term toxicity | Until death of the patients
Evaluation of QoL | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FEUGIER, MD, Principal Investigator — CHU Brabois, 54511 Vandoeuvre les Nancy
Locations (116):
- Belgium (24):
  - ZNA Stuivenberg, Antwerp
  - Clinique Sud du Luxembourg, Arlon
  - RHMS, Baudour
  - A. Z. Sint-Jan, Bruges
  - CHU Brugmann, Brussels
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - Université Catholique de Louvain Saint Luc, Brussels
  - CH Notre Dame, Charleroi
  - CHU Charleroi-Vésale, Charleroi
  - Centre de Santé des Fagnes, Chimay
  - Clinique Notre Dame de Grace, Gosselies
  - Hôpital Jolimont, Haine-Saint-Paul
  - CH Hutois, Huy
  - AZ Groeninge - Campus Maria's Voorzienigheid, Kortrljk
  - CHU Tivoli, La Louvière
  - CHR de la Citadelle, Liège
  - CHU de Liège, Liège
  - CHU Ambroise Paré, Mons
  - Clinique Saint Joseph, Mons
  - Hôpital Sainte Elisabeth, Namur
  - Heilig Hart Ziekenhuis, Roeselare
  - Centre Hospitalier de Wallonie Picarde - CHwapi, Tournai
  - CH de la Tourelle-Peltzer, Verviers
  - UCL Mt Godinne, Yvoir
- France (92):
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU Amiens - Hôpital Sud, Amiens
  - CHU d'Angers, Angers
  - CH Antibes, Antibes
  - CH Victor Dupouy, Argenteuil
  - CH d'Avignon - Hôpital Henri Dufaut, Avignon
  - Hôpital de Bayonne, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - CH Jean Minjoz, Besançon
  - CH Béziers, Béziers
  - Centre Hospitalier de Blois, Blois
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH Dr Duchenne, Boulogne-sur-Mer
  - CH de Bourg en Bresse, Bourg-en-Bresse
  - CHU Morvan, Brest
  - Centre Hospitalier de Brive, Brive-la-Gaillarde
  - CHU Clémenceau, Caen
  - Centre Francois Baclesse, Caen
  - CH Cannes, Cannes
  - CH Chambéry, Chambéry
  - CH de Chartres, Chartres
  - Hôpital de Châlon, Châlon Sur Saône
  - Hôpital Antoine Béclère, Clamart
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Pôle Santé Publique, Clermont-Ferrand
  - CH de Compiègne, Compiègne
  - Hôpital Sud Francilien, Corbeil Essonne
  - Hôpital Henri Mondor, Créteil
  - CHU le Bocage, Dijon
  - CH de Dunkerque, Dunkirk
  - CH Fréjus St Raphaël, Fréjus
  - CHU Grenoble, Grenoble
  - Centre Hospitalier de Guéret, Guéret
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Laval, Laval
  - Hôpital André Mignot, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU LIMOGES - Hôpital Universitaire Dupuytren, Limoges
  - CH de Bretagne Sud, Lorient
  - Clinique de la Sauvegarde, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH les Chanaux, Mâcon
  - CH de Meaux, Meaux
  - Ch Marc Jacquet, Melun
  - Hôpital Notre Dame de Bon Secours, Metz
  - CH Saint-Eloi, Montpellier
  - CRCL Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - CHU de Mulhouse - Hôpital Emile Muller, Mulhouse
  - Centre Catherine de Sienne, Nantes
  - CHU Hôtel Dieu, Nantes
  - Hôpital Américain de Paris, Neuilly
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - CHU Caremeau, Nîmes
  - Clinique Valdegour, Nîmes
  - CHR de la Source, Orléans
  - Hôpital Saint Antoine, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Necker, Paris
  - Hôpital Hôtel Dieu, Paris
  - Institut Curie, Paris
  - Hôpital St Louis, Paris
  - CH Saint Jean, Perpignan
  - Hôpital Haut Levêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - CH René Dubos, Pontoise
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - Hôpital Robert Debré, Reims
  - Clinique de Courlancy, Reims
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Mathilde, Rouen
  - CHU Saint-Etienne, Saint Priest En Jarest
  - Centre René Huguenin, Saint-Cloud
  - CHG St Germain, Saint-Germain-en-Laye
  - CH de Saint Quentin, Saint-Quentin
  - CHU de Saint Malo, St-Malo
  - Hôpital Font Pré, Toulon
  - CHU Bretonneau, Tours
  - Hôpital de Troyes, Troyes
  - CH de Valence, Valence
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Gyan E, Sonet A, Brice P, Anglaret B, Laribi K, Fruchart C, Tilly H, Araujo C, Soubeyran P, Gonzalez H, Morineau N, Nicolas-Virelizier E, Ghesquieres H, Salles B, Bouabdallah R, Orfeuvre H, Fahri J, Couturier O, Xerri L, Feugier P; Lymphoma Study Association (LYSA). Bendamustine and rituximab in elderly patients with low-tumour burden follicular lymphoma. Results of the LYSA phase II BRIEF study. Br J Haematol. 2018 Oct;183(1):76-86. doi: 10.1111/bjh.15513. Epub 2018 Aug 16. PMID 30117149